CLINICAL TRIAL: NCT03677817
Title: Prospective, Randomized, Double Blind, Superiority Trial, Evaluating the Effect of Perioperative Lidocaine on Postoperative Opioid Consumption, Pain Ratings, Duration of Hospital Stay, Time to First Defecation, 30-day Mortality and Development of Chronic Pain in Patients Undergoing Video-assisted Thoracoscopic Procedures
Brief Title: Perioperative Lidocaine Administration in Thoracoscopic Surgery for Improved Postoperative Pain Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-00259; ch15Toffel
Record Dates: First submitted 2018-09-11; First posted 2018-09-19 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Postoperative Pain
Keywords: thoracoscopic surgery; Perioperative intravenous lidocaine administration; Lidocaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): perioperative IV administration regimen of lidocaine will be as follows: 1.5 mg/kg IV induction bolus dose (before intubation and at least 30 minutes before incision) followed by continuous infusion of 3.mg/kg/h, until 2 hours after skin closure
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): perioperative IV administration regimen of placebo solution (NaCl 0,9%) will be as follows: induction bolus (before intubation and at least 30 minutes before incision) followed by continuous infusion of placebo solution (NaCl 0,9%) until 2 hours after skin closure
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: Lidocaine — regimen of lidocaine administration of 1,5 mg/kg, IV bolus, followed by continuous infusion at 3,0 mg/kg/h
  Arms: Lidocaine
Drug: NaCl 0,9% — IV bolus of NaCl 0,9%, followed by continuous infusion of NaCl 0,9%
  Arms: Placebo

SUMMARY:
Placebo-controlled study to analyze the effect of perioperative intravenous lidocaine administration on total morphine consumption (TMC) and on pain intensity in thoracoscopic surgery .

DETAILED DESCRIPTION:
Thoracoscopy (thoracic surgery) is a video-assisted minimally invasive operation in thoracic surgery, which is associated with pain after surgery. Trial drug Lidocaine is approved as pain medication. This placebo-controlled study analyzes the effect of perioperative intravenous lidocaine administration on total morphine consumption (TMC) and on pain intensity in thoracoscopic surgery .

Half of the patients will receive NaCl 0.9% (a saline solution without active ingredient) instead of Lidocaine.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing video-assisted thoracoscopic procedures under general anaesthesia.
* American Society of Anesthesiologists (ASA) physical Status classes I to III
* age ≥ 18 years
* Patient informed consent

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product
* Contraindications to self-administration of opioids
* Women who are pregnant or breast feeding
* Steroid therapy
* Chronic pain therapy
* Atrioventricular block grade II to III
* Congestive heart failure
* Liver insufficiency
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Change in total morphine consumption (TMC) | within the first 24 hours, measured at 1 hour, 2 hours, 4 hours, 8 hours, 16 hours, and 24 hours after skin closure
  change in total morphine consumption (TMC) via Patient Controlled Analgesia (PCA)
change in pain intensity | within the first 24 hours, measured at 1 hour, 2 hours, 4 hours, 8 hours, 16 hours, and 24 hours after skin closure
  change in pain intensity of at least 1.5 units on the Visual Analogue Scale (VAS). The pain VAS is a unidimensional measure of pain intensity; the scale is anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale])

SECONDARY OUTCOMES:
Duration of hospital stay | from day of surgery until day of discharge from hospital (an average of 2 days)
  length of hospital stay (in days)
time to first defecation - Defined as the time from skin closure to the time of first defecation | From timepoint of surgical skin closure (end of surgery) to the timepoint of first defecation after surgical skin closure (an average of 2 days)
  time to first defecation - Defined as the time from skin closure to the time of time to first defecation (measured in hours)
Change in chronic pain | 2 weeks, 3 months and 6 months after surgery
  Change in pain intensity (with and without coughing) on the Visual Analogue Scale (VAS). The pain VAS is a unidimensional measure of pain intensity; the scale is anchored by "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale])
occurrence of nausea and/or vomiting | from the date of surgery until the date of discharge from hospital (an average of 2 days)
  occurrence of nausea and/or vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Didier Lardinois, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Division of Thoracic Surgery,University Hospital of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Hojski A, Bolliger D, Mallaev M, Dackam S, Tsvetkov N, Wiese M, Schneider T, Lampart A, Lardinois D. Perioperative intravenous lidocaine in thoracoscopic surgery for improved postoperative pain control: a randomized, placebo-controlled, double-blind, superiority trial. J Thorac Dis. 2024 Mar 29;16(3):1923-1932. doi: 10.21037/jtd-23-1438. Epub 2024 Mar 25. PMID 38617784